CLINICAL TRIAL: NCT02558959
Title: Effect of Second-line Irinotecan and Capecitabine Versus Irinotecan Alone in Advanced Biliary Tract Cancer Patients Progressed After First-line Gemcitabine and Cisplatin: A Randomized Controlled Study
Brief Title: Second-line Irinotecan and Capecitabine Versus Irinotecan for Gemcitabine and Cisplatin Refractory Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, Director of Cancer Biotherapy Center, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZYYYMedOncoBIL01
Record Dates: First submitted 2015-09-21; First posted 2015-09-24 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Biliary Tract Neoplasms
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Irinotecan; Capecitabine

ARMS (2):
- Irinotecan and Capecitabine (Experimental): irinotecan 180mg/m2 d1, capecitabine 1000mg/m2 bid d1-10, q2w
  Interventions: Drug: Irinotecan; Drug: Capecitabine
- Irinotecan (Active Comparator): irinotecan 180mg/m2 d1, q2w
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan
Drug: Capecitabine
  Arms: Irinotecan and Capecitabine

SUMMARY:
This study is designed to investigate the effect of second-line irinotecan and capecitabine versus irinotecan alone for gemcitabine and cisplatin refractory advanced biliary tract cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed advanced biliary tract cancer who had experienced progression during first-line gemcitabine and cisplatin
* Age 18 years or older
* Measurable reference cancer site(s) confirmed with computed tomography (CT) or magnetic resonance imaging (MRI)
* Karnofsky performance status (KPS) of at least 70%
* Adequate renal function, adequate hepatic function, adequate bone marrow function

Exclusion Criteria:

* The presence of any severe concomitant disease that could interrupt the planned treatment
* Intractable pain
* Hypersensitivity to study drugs
* Serious cardiovascular disease
* If female, pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | within 1 year
  PFS

SECONDARY OUTCOMES:
Overall Survival | within 1 year
  OS

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China